CLINICAL TRIAL: NCT00974194
Title: Single Port vs Tree Trocars Laparoscopic Cholecystectomy: a Randomized Controlled Trial
Brief Title: Safety and Cost-effectiveness Study of Single Port Laparoscopic Cholecystectomies
Acronym: SPoCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, professor of surgery, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPoCOT_2009
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Cholecystolithiasis
Keywords: Cholecystolithiasis; Cholecystectomy; Laparoscopic surgery; Single port
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SinglePort CCK (Experimental): CCK using Triport
  Interventions: Procedure: Single Trocar CCK
- LS CCK (Active Comparator): CCK using three or four trocars
  Interventions: Procedure: Standard CCK

INTERVENTIONS:
Procedure: Single Trocar CCK — CCK using Triport
  Arms: SinglePort CCK
Procedure: Standard CCK — CCK using three or four ports
  Arms: LS CCK

SUMMARY:
Many feasibility studies have been published on Single Port surgery, but no comparative studies have shown any advantages compared to standard laparoscopy. The purpose of this study is to compare the clinical outcomes and economical issues of laparoscopic cholecystectomies using single port transumbilical approach and three trocars.

DETAILED DESCRIPTION:
Design:

* Prospective Randomized Controlled trial
* Population analysis based on Intention To Treat
* Patient and data analyzer blinded (double-blind trial)

Outcomes observed:

* Primary: pain
* Secondaries: overall operative time, complication rate, cost-effectiveness analysis, cosmetic evaluation, quality of life, CO2 consumption

Nbr of patients included: 260

Port used: Triport, Olympus

ELIGIBILITY:
Inclusion Criteria:

* Cholecystolithiasis
* Age 18 to 75 y.o.
* BMI < 35

Exclusion Criteria:

* Immunodeficiency
* Choledocholithiasis
* Previous upperGI open surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Pain (value on a Visual Analog Scale) | 1 day
  VAS
Pain (value on a Visual Analog Scale) | 2 days
  VAS
Pain (value on a Visual Analog Scale) | 1 month
  VAS
Pain (value on a Visual Analog Scale) | 3 month
  VAS
Pain (value on a Visual Analog Scale) | 1 year
  VAS

SECONDARY OUTCOMES:
Complications | 1 month
  In euro
Operative time | Operative day
  In euro
Cost analysis | 1 year
  In euro
Cosmetic results | 1 month
  According to POSAS score
Cosmetic results | 3 month
  According to POSAS score
Cosmetic results | 1 year
  According to POSAS score
Complications | 3 month
  According to Clavien classification and CCI
Complications | 1 year
  According to Clavien classification and CCI

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Allemann, MD, Principal Investigator — CHV/CHUV
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland

REFERENCES:
- See also: Internet page of our departement — http://www.chirurgieviscerale.ch